CLINICAL TRIAL: NCT07364188
Title: Bronchodilator Response in COPD and Asthma: Correlation Between Spirometry, IOS Indices, and Dyspnea Relief
Status: Not yet recruiting | Type: Observational
Sponsor: Allergi- og Lungeklinikken, Elsinore (Network)
Responsible Party: Sponsor
Other Study IDs: F-25059703
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Asthma Bronchiale; COPD; Bronchodilation; Spirometry; Impedance; Small Airways Disease
Keywords: asthma; COPD; Correlation; Bronchodilator response; MCID
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma: FEV1/Forced Vital Capacity (FVC) <0.7 at baseline (7) Visual Analog Scale (VAS) dyspnea score ≥10 (0-100, 100 max) (25,26). Doctor diagnosed asthma Less than 10 packyears.
  Exclusion Criteria:
  * Patients aged less than 18 years old.
  * Not able to perform spirometry or impulse oscillometry.
  * Cognitive disorders and not able to answer Asthma Control Questionnaire (ACQ), VAS dyspnea score, and COPD Assessment Test (CAT) score (25-28).
  * Short-acting beta-agonists 6 h, long-acting beta-agonists 2 days, short-acting anti-muscarinic agent 12 h, Long-acting anti-muscarinic agents 2 days.
  * Comorbidities with significant influence on dyspnea eg. bronchiectasis, ILS, mb. Cordis, lung resection, anemia, and active malignant disease
  * BMI ≥40 kg/m2.
  Interventions: Diagnostic Test: Bronchodilator
- COPD: FEV1/Forced Vital Capacity (FVC) <0.7 at baseline (7) Visual Analog Scale (VAS) dyspnea score ≥10 (0-100, 100 max) (25,26).
  Doctor diagnosed COPD Smokers or ex-smokers with ≥10 packyears
  Exclusion Criteria:
  * Patients aged less than 18 years old.
  * Not able to perform spirometry or impulse oscillometry.
  * Cognitive disorders and not able to answer Asthma Control Questionnaire (ACQ), VAS dyspnea score, and COPD Assessment Test (CAT) score (25-28).
  * Short-acting beta-agonists 6 h, long-acting beta-agonists 2 days, short-acting anti-muscarinic agent 12 h, Long-acting anti-muscarinic agents 2 days.
  * Comorbidities with significant influence on dyspnea eg. bronchiectasis, ILS, mb. Cordis, lung resection, anemia, and active malignant disease
  * BMI ≥40 kg/m2.
  Interventions: Diagnostic Test: Bronchodilator

INTERVENTIONS:
Diagnostic Test: Bronchodilator — Classic beta-2-reversibility test

SUMMARY:
A bronchodilator reversibility test is widely used in the diagnosis and management of obstructive lung diseases.

Bronchodilators relieve symptoms in asthma and COPD. Traditionally, their effectiveness has been assessed using spirometric indices, particularly FEV₁. However, changes in FEV₁ often do not correlate well with patients' subjective experience of dyspnoea relief or with changes in small airway function.

Impulse oscillometry (IOS) provides an effort-independent assessment of respiratory mechanics during tidal breathing and is more sensitive to small airway dysfunction than spirometry. Despite this, the clinical utility of IOS in routine COPD and asthma assessment remains underexplored, and its relationship to both spirometric response and symptom relief is not fully established, and the Minimal Clinically Important Difference (MCID) for IOS parameters has not been firmly established. Determining the MCID is essential for interpreting individual patient responses in a clinically meaningful way and for guiding treatment decisions in both research and practice.

Hypothesis & Aims

In patients with either asthma or COPD baseline values and bronchodilator responses are compared. More specifically, this study aims to:

1. assess baseline correlations: Evaluate the correlation between ΔX5-baseline (EFL expiratory flow limitation=small airway collapse during expiration), RV/TLC-baseline, X5-average at baseline, FEV1-baseline, VAS-dyspnea at baseline, and ACQ-6-baseline.
2. compare bronchodilator responses across methods: Examine the correlation between bronchodilator-induced changes in FEV₁ and IOS parameters (including both average and delta values) and explore their relationship with short-term changes in dyspnea.
3. establish clinical relevance: Determine the MCID for key IOS variables using both anchor-based and distribution-based approaches, anchored to perceived changes in lung symptoms.

DETAILED DESCRIPTION:
Introduction and aims: see brief summary.

Method and Patients This is a real-life, cross-sectional analysis of a single-centered, observational study on 60 adult patients with clinical diagnosed asthma and 60 COPD patients, consecutively recruited between February 1, 2026, and June 30, 2027, and followed at least 6 months for diagnostic clarification.

Inclusion Criteria:

Both asthma and COPD patients:

1. Written informed consent.
2. FEV1/Forced Vital Capacity (FVC) <0.7 at baseline )
3. Visual Analog Scale (VAS) dyspnea score ≥10 (0-100, 100 max).

Asthma: Doctor diagnosed asthma 1. less than 10 packyears.

COPD: Doctor diagnosed COPD with FEV1/FVC <0.7 post-bronchodilation

1. Smokers or ex-smokers with ≥10 packyears

Exclusion Criteria:

* Patients aged less than 18 years old.
* Not able to perform spirometry or impulse oscillometry.
* Cognitive disorders and not able to answer Asthma Control Questionnaire (ACQ), VAS dyspnea score, and COPD Assessment Test (CAT) score.
* Short-acting beta-agonists 6 h, long-acting beta-agonists 2 days, short-acting anti-muscarinic agent 12 h, Long-acting anti-muscarinic agents 2 days.
* Comorbidities with significant influence on dyspnea eg. bronchiectasis, ILS, mb. Cordis, lung resection, anemia, and active malignant disease
* BMI ≥40 kg/m2.

It is a real-life study where most patients are followed up within 6 months. The diagnosis - asthma, COPD, or other condition - may change after follow-up (maximum 6 months after the index examination).

Minimal Clinical Important Difference

Anchor-Based Methods:

1. The receiver operating characteristic (ROC) curve-based method determines the minimum clinically important difference (MCID) by identifying the value that maximizes the Youden Index. This index is calculated as the maximum sum of sensitivity and specificity. Using data from patients who rate themselves "a little better" and patients who rate themselves "no change"
2. The social comparison approach provides the MCID as the mean of two differences: the difference of mean score between patients who rate themselves as "a little worse" and patients who rate themselves "no change".
3. Within-patients score change MCID is the mean delta score of patients who rate themselves "a little better".
4. The methods of 95% limits of upper agreement: MCID is the mean delta score -1.96 standard error of the delta score of the patients who answered "no change"

Distribution-Based Methods:

1. MCID defined as standard error of measurement (SEM) evaluated on the baseline values from patients who rated themselves "no change".
2. MCID defined as 0.5 SD of delta score from patients who answered "a little better"
3. MCID is defined as 1.96 × √2 × SEM, assessed on baseline values from patients who reported "no change", which represents the smallest change in a measurement that can be considered a "real" change, rather than just random measurement error.

Brochodilator test and order of test To avoid or minimize the effect of deep inhalation on IOS, IOS was performed at least 15 minutes after spirometry and body box.

Patients were administered 4 doses of 0.1 mg Ventoline (salbutamol) via pressurized metered-dose inhaler and spacer (Aero Champer). Post-IOS and post-spirometry were performed 15-20 minutes after the bronchodilator inhalation

ELIGIBILITY:
Inclusion Criteria:

* Both asthma and COPD patients:

  1. Written informed consent.
  2. FEV1/Forced Vital Capacity (FVC) <0.7 at baseline (7)
  3. Visual Analog Scale (VAS) dyspnea score ≥10 (0-100, 100 max) (25,26).
* Asthma: Doctor diagnosed asthma

  1. less than 10 packyears.
* COPD: Doctor diagnosed COPD with FEV1/FVC <0.7 post-bronchodilation 1. Smokers or ex-smokers with ≥10 packyears

Exclusion Criteria:

* Patients aged less than 18 years old.
* Not able to perform spirometry or impulse oscillometry.
* Cognitive disorders and not able to answer Asthma Control Questionnaire (ACQ), VAS dyspnea score, and COPD Assessment Test (CAT) score (25-28).
* Short-acting beta-agonists 6 h, long-acting beta-agonists 2 days, short-acting anti-muscarinic agent 12 h, Long-acting anti-muscarinic agents 2 days.
* Comorbidities with significant influence on dyspnea eg. bronchiectasis, ILS, mb. Cordis, lung resection, anemia, and active malignant disease
* BMI ≥40 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: referred to Allergy and Lung Clinic Elsinore, Denmark for evaluation of Asthma and COPD (obstructive lung disease)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
FEV1 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Forced expiratory volumen in one second, L and % predicted
X5 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Reactance at 5 Hz; kPa/L/s
Dyspnoea | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Visual analog scale (0-100); 0 means no dyspnoea, and 100 means maximum dyspnoea

SECONDARY OUTCOMES:
R5 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Resistance at 5 Hz, kPa/L/s and % predicted
R5-R20 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Resistance in small airways, kPa/L/s
Fres | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Resonant frequency (stiffness), Hz
AX | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Area of reactance, kPa/L
Delta-X5 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Inspiratory - expiratory difference in X5, kPa/L/s
Delta R5 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Inspiratory - expiratory difference in R5 (total resitance), kPa/L/s
FEF 25-75 | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  Expiratory Flow at 25% to 75% during spirometry, L and % predicted
FEV1/FVC-ratio | Before and 20 minuttes after inhaled Salbutamol 0.4 mg
  FEV1/forced expiratory capacity (FVC)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Ringbæk, MSci, Principal Investigator — Allergi og Lungeklinikken Helsingør

IPD SHARING:
Plan to Share IPD: No
I have not applied for permission to share data with others.

REFERENCES:
- [Background] Szalai AJ, van Ginkel FW, Wang Y, McGhee JR, Volanakis JE. Complement-dependent acute-phase expression of C-reactive protein and serum amyloid P-component. J Immunol. 2000 Jul 15;165(2):1030-5. doi: 10.4049/jimmunol.165.2.1030. PMID 10878380
- [Background] Proskurov VA. [Prevention of staph infections in maternity hospitals]. Pediatriia. 1969 Nov;48(11):49-52. No abstract available. Russian. PMID 5392482
- [Background] Dean J, Kolsum U, Hitchen P, Gupta V, Singh D. Clinical characteristics of COPD patients with tidal expiratory flow limitation. Int J Chron Obstruct Pulmon Dis. 2017 May 22;12:1503-1506. doi: 10.2147/COPD.S137865. eCollection 2017. PMID 28579768
- [Background] Paredi P, Goldman M, Alamen A, Ausin P, Usmani OS, Pride NB, Barnes PJ. Comparison of inspiratory and expiratory resistance and reactance in patients with asthma and chronic obstructive pulmonary disease. Thorax. 2010 Mar;65(3):263-7. doi: 10.1136/thx.2009.120790. PMID 20335298
- [Background] Bloom DA, Kaplan DJ, Mojica E, Strauss EJ, Gonzalez-Lomas G, Campbell KA, Alaia MJ, Jazrawi LM. The Minimal Clinically Important Difference: A Review of Clinical Significance. Am J Sports Med. 2023 Feb;51(2):520-524. doi: 10.1177/03635465211053869. Epub 2021 Dec 2. PMID 34854345
- [Background] Saadeh C, Saadeh C, Cross B, Gaylor M, Griffith M. Advantage of impulse oscillometry over spirometry to diagnose chronic obstructive pulmonary disease and monitor pulmonary responses to bronchodilators: An observational study. SAGE Open Med. 2015 Apr 6;3:2050312115578957. doi: 10.1177/2050312115578957. eCollection 2015. PMID 26770777
- [Background] Cottee AM, Seccombe LM, Thamrin C, King GG, Peters MJ, Farah CS. Bronchodilator Response Assessed by the Forced Oscillation Technique Identifies Poor Asthma Control With Greater Sensitivity Than Spirometry. Chest. 2020 Jun;157(6):1435-1441. doi: 10.1016/j.chest.2019.12.035. Epub 2020 Jan 23. PMID 31982392
- [Background] Greig R, Stewart K, Chan R, Lipworth B. Assessment of bronchodilator responsiveness using low-frequency impedance in type 2-high uncontrolled severe asthma. Ann Allergy Asthma Immunol. 2025 Feb;134(2):231-232. doi: 10.1016/j.anai.2024.10.011. Epub 2024 Oct 9. No abstract available. PMID 39383941
- [Background] Kaminsky DA, Simpson SJ, Berger KI, Calverley P, de Melo PL, Dandurand R, Dellaca RL, Farah CS, Farre R, Hall GL, Ioan I, Irvin CG, Kaczka DW, King GG, Kurosawa H, Lombardi E, Maksym GN, Marchal F, Oostveen E, Oppenheimer BW, Robinson PD, van den Berge M, Thamrin C. Clinical significance and applications of oscillometry. Eur Respir Rev. 2022 Feb 9;31(163):210208. doi: 10.1183/16000617.0208-2021. Print 2022 Mar 31. PMID 35140105
- [Background] King GG, Bates J, Berger KI, Calverley P, de Melo PL, Dellaca RL, Farre R, Hall GL, Ioan I, Irvin CG, Kaczka DW, Kaminsky DA, Kurosawa H, Lombardi E, Maksym GN, Marchal F, Oppenheimer BW, Simpson SJ, Thamrin C, van den Berge M, Oostveen E. Technical standards for respiratory oscillometry. Eur Respir J. 2020 Feb 27;55(2):1900753. doi: 10.1183/13993003.00753-2019. Print 2020 Feb. PMID 31772002
- [Background] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213
- [Background] Janson C, Malinovschi A, Amaral AFS, Accordini S, Bousquet J, Buist AS, Canonica GW, Dahlen B, Garcia-Aymerich J, Gnatiuc L, Kowalski ML, Patel J, Tan W, Toren K, Zuberbier T, Burney P, Jarvis D. Bronchodilator reversibility in asthma and COPD: findings from three large population studies. Eur Respir J. 2019 Sep 5;54(3):1900561. doi: 10.1183/13993003.00561-2019. Print 2019 Sep. PMID 31221806
- [Background] Kaminsky DA. What Is a Significant Bronchodilator Response? Ann Am Thorac Soc. 2019 Dec;16(12):1495-1497. doi: 10.1513/AnnalsATS.201908-604ED. No abstract available. PMID 31774318
- [Background] Beasley R, Hughes R, Agusti A, Calverley P, Chipps B, Del Olmo R, Papi A, Price D, Reddel H, Mullerova H, Rapsomaniki E. Prevalence, Diagnostic Utility and Associated Characteristics of Bronchodilator Responsiveness. Am J Respir Crit Care Med. 2024 Feb 15;209(4):390-401. doi: 10.1164/rccm.202308-1436OC. PMID 38029294
- [Background] Chan R, Lipworth BJ. Oscillometry bronchodilator response in adult moderate to severe eosinophilic asthma patients: A prospective cohort study. Clin Exp Allergy. 2022 Sep;52(9):1118-1120. doi: 10.1111/cea.14185. Epub 2022 Jun 22. No abstract available. PMID 35707948